CLINICAL TRIAL: NCT01980680
Title: The Exogenous Progesterone Free Luteal Phase After GnRHa Trigger - a Randomized Controlled Pilot Study in Normo-responder IVF Patients
Brief Title: The Exogenous Progesterone Free Luteal Phase After GnRHa Trigger - a Pilot Study in Normo-responder IVF Patients
Acronym: GnRHa trigger
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peter Humaidan (Other)
Responsible Party: Sponsor-Investigator, Peter Humaidan, Professor, Regionshospitalet Viborg, Skive
Organization: Regionshospitalet Viborg, Skive (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Agonist5
Record Dates: First submitted 2013-10-28; First posted 2013-11-11 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Progesterone; Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Agonist trigger (Experimental): Agonist trigger Buserelin 0,5 mg and Pregnyl (hCG)
  Interventions: Drug: hCG
- hCG (Active Comparator): hCG trigger Pregnyl (hCG) and Progesterone and Estradiol
  Interventions: Drug: Progesterone and Estradiol

INTERVENTIONS:
Drug: hCG
  Arms: Agonist trigger
Drug: Progesterone and Estradiol
  Arms: hCG

SUMMARY:
After hCG trigger a large amount of exogenous progesterone is used for luteal phase support in many countries until 10th week of gestation. Instead we suggest the use of two small doses of hCG after the trigger during the early luteal phase after GnRHa trigger, promoting the endogenous progesterone production from the corpora lutea (CL).

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 40
* Normal menstrual cycles: 25-34 days
* Oligomenorrhea/amenorrhea or polycystic syndrome (defined according to the Rotterdam criteria 2004)
* BMI >18 and <35 kg/m2

Exclusion Criteria:

* Patients with >14 follicles on day of trigger
* Previous hyperresponse with OHSS development
* Previous low response (less than 3 oocytes on a high dose of FSH stimulation)
* Endocrine disorders

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-12; Primary Completion 2019-09 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate per patient | 10th week of gestation.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fertility Clinic, Regional Hospital of Skive, Skive, Denmark